CLINICAL TRIAL: NCT00771316
Title: A Phase 3, Randomized, Active Comparator-Controlled Clinical Trial to Study the Safety and Efficacy of MK0826 and Meropenem in Patients With Complicated Urinary Tract Infection
Brief Title: Clinical Trial to Study the Safety and Effectiveness of MK0826 and Other Antibiotic Therapy in Patients With Complicated Urinary Tract Infection (0826-054)
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: feasibility and low enrollment
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0826-054; MK0826-054; 2008_562
Record Dates: First submitted 2008-10-09; First posted 2008-10-13 (Estimated); Results first posted 2010-07-09 (Estimated); Last update posted 2017-03-21 (Actual); Status verified 2017-02

CONDITIONS: Urinary Tract Infections
MeSH Terms: conditions — Urinary Tract Infections | interventions — Ertapenem

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- Group 1 (Experimental): MK0826 (ertapenem)
  Interventions: Drug: MK0826 (ertapenem)
- Group 2 (Active Comparator): meropenem
  Interventions: Drug: Comparator: meropenem

INTERVENTIONS:
Drug: MK0826 (ertapenem) — A single dose of 1.0g IV infused over a 30 minute interval at hour 0
  Arms: Group 1
Drug: Comparator: meropenem — 500 mg IV infused over a 30 minute interval at hours 0, 8, and 16 for at least 4 days
  Arms: Group 2

SUMMARY:
The purpose of this study is to demonstrate that MK0826 is comparable to Meropenem in the treatment of complicated Urinary Tract Infections (UTIs) in adults.

ELIGIBILITY:
Inclusion Criteria:

* Patient has a clinically suspected and /or bacteriologically documented complicated UTI or acute pyelonephritis judged by the investigator to be serious
* Patient has one positive urine culture within 48 hours of enrollment
* Patient has one or more signs or symptoms of either upper or lower UTI
* Patient is male with or without a bladder catheter or urologic abnormalities; OR patient is a female with a history or clinical evidence of one or more urologic abnormalities

Exclusion Criteria:

* Patient has received any amount of effective concomitant antibiotic therapy after obtaining the urine culture for admission to this study (admission urine culture) and prior to the administration of the first dose of study antibiotics
* Patient's infection has been treated with greater than 24 hours of systemic antibiotic therapy known to be effective against the presumed or documented pathogens within the 72 hour period immediately prior to consideration for entry into the study
* Patient has complete obstruction of any portion of the urinary tract. Patient has a history of seizures other than an uncomplicated febrile seizure

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2008-12; Primary Completion 2009-06 (Actual); Study Completion 2009-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: Yes
http://www.merck.com/clinical-trials/pdf/Merck%20Procedure%20on%20Clinical%20Trial%20Data%20Access%20Final_Updated%20July_9_2014.pdf
  http://engagezone.msd.com/ds_documentation.php

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Phase III
  First patient enrolled on 09-Dec-2008
  Last patient enrolled on 12-May-2009
  The last patient's last visit was 08-Jun-2009
  The study was conducted at 6 study centers in the United States and Europe.
  Study was terminated early due to feasibility issues including slow enrollment.
Groups:
- MK0826 (Ertapenem): MK0826-Patient received a once daily, intravenous infusion of 1.0g of MK0826 plus placebo (0.9% saline) at Hours 0, 8 and 16 for at least 4 days.
- Meropenem: Meropenem-Patient received a once daily, intravenous infusion of 500 mg of meropenem at Hours 0, 8 and 16 for at least 4 days.
Period: Overall Study
Arm/Group | MK0826 (Ertapenem) | Meropenem
Started | 4 | 2
Completed | 2 | 1
Not Completed | 2 | 1
Not completed — Adverse Event | 0 | 1
Not completed — Patient withdrew consent | 1 | 0
Not completed — Discontinued due to early termination | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | MK0826 (Ertapenem) | Meropenem | Total
Number analyzed (Participants) | 4 | 2 | 6
Age, Continuous [Mean (Full Range); unit: years] | 37.75 [21 to 50] | 58 [58 to 58] | 44.5 [21 to 58]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 0 | 2
  Male | 2 | 2 | 4
Race/Ethnicity, Customized [Number; unit: participants]
  White | 4 | 2 | 6

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Serious Urinary Tract Infection With an Overall Microbiological Response to MK0826 Compared to Meropenem at the 5 to 9 Day Post Therapy Early Follow-up Visit
Description: Microbiological response defined as: 1) Eradication-urine culture shows reduced uropathogen, 2)Persistence-urine culture taken after at least 2 days of therapy grows the original uropathogen, 3)Persistence with Acquisition of Resistance- urine culture taken after at least 2 days of therapy grows the original uropathogen but shows resistance to study drug, 4)Superinfection-Growth of uropathogen other than original pathogen, 5)New Infection-A new pathogen grows other than the original uropathogen, 6)Indeterminate-Any circumstance where impossible to define microbiological response.
Time Frame: 5 to 9 days post therapy
Population: This analysis was not completed due to early termination of the study.
Arm/Group | MK0826 (Ertapenem) | Meropenem
Number analyzed (Participants) | 0 | 0

2. Primary Outcome: Number of Participants With Serious Urinary Tract Infection With a Clinical Response to MK0826 Compared to Meropenem at Discontinuation of Intravenous Therapy (DCIV)
Description: Clinical response at DCIV defined as: 1) Improved-All or most pretherapy signs and symptoms of infection have improved and no additional antibiotic is required, 2) Failure-No response to therapy, persistence or progression of pretherapy signs and symptoms, 3) Indeterminate-Study data not available due to complications related to underlying medical condition, patient withdrawn from study or extenuating circumstances preclude classification as improved or failure.
Time Frame: After at least 4 days of IV therapy
Population: This analysis was not completed due to early termination of the study.
Arm/Group | MK0826 (Ertapenem) | Meropenem
Number analyzed (Participants) | 0 | 0

3. Primary Outcome: Number of Participants With Serious Urinary Tract Infection With an Overall Microbiological Response to MK0826 Compared to Meropenem at Discontinuation of Intravenous Therapy (DCIV)
Description: as for outcome 1
Time Frame: After at least 4 days of IV therapy
Population: This analysis was not completed due to early termination of the study.
Arm/Group | MK0826 (Ertapenem) | Meropenem
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Any serious adverse experience, including death due to any cause, which occurred to any subject entered in the study or within 14 days following cessation of treatment.
Arm/Group | MK0826 (Ertapenem) | Meropenem
Serious Adverse Events (participants affected / at risk) | 0/4 | 1/2
Other Adverse Events (participants affected / at risk) | 1/4 | 0/2
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | MK0826 (Ertapenem) (N=4) | Meropenem (N=2)
Shortness of breath (General disorders) | 0 | 1
Chest pain (General disorders) | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | MK0826 (Ertapenem) (N=4) | Meropenem (N=2)
Mouth dryness (Gastrointestinal disorders) | 1 | 0

LIMITATIONS AND CAVEATS:
The reason for early termination: Study was terminated early due to feasibility issues including slow enrollment.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Merck agreements may vary with individual investigators, but will not prohibit any investigator from publishing. Merck supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.